CLINICAL TRIAL: NCT02629991
Title: Oxytocin vs. Placebo for the Treatment Hyperphagia in Children and Adolescents With Prader-Willi Syndrome
Acronym: OXT-PWS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Principal Investigator, Eric Hollander, Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-10-427-01
Record Dates: First submitted 2015-10-18; First posted 2015-12-15 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Prader-Willi Syndrome; Hyperphagia
Keywords: Prader-Willi Syndrome (PWS); Hyperphagia
MeSH Terms: conditions — Prader-Willi Syndrome; Hyperphagia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Oxytocin (Experimental): Participants were instructed to take 16 IU/per day everyday (2 puffs per nostril, 4 IU each puff).
  Interventions: Drug: Intranasal Oxytocin (IN-OXT)
- Matched Placebo (Placebo Comparator): Participants were instructed to take 16 IU/per day everyday (2 puffs per nostril, 4 IU each puff).
  Interventions: Other: Matched Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin (IN-OXT) — Participants were instructed to take 16 IU/per day everyday (2 puffs per nostril, 4 IU each puff).
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Other: Matched Placebo — Participants were instructed to take 16 IU/per day everyday (2 puffs per nostril, 4 IU each puff).
  Arms: Matched Placebo

SUMMARY:
The investigators propose a randomized double-blind 8 week treatment trial of intranasal oxytocin (IN-OXT) vs. placebo in 24 subjects aged 5 to 18 years with PWS in order to assess IN-OXT's affect on (1) Eating behaviors (2) Repetitive and disruptive behaviors and (3) Salivary OXT levels.

DETAILED DESCRIPTION:
The investigators propose to conduct a treatment study of intranasal oxytocin (IN-OXT) vs. placebo in children and adolescents with Prader-Willi Syndrome (PWS). OXT has already been proven safe and effective in a treatment study of socialization and disruptive behavior in adults with PWS and is being used in infants with PWS in an ongoing clinical trial. The investigators hypothesize that OXT will be superior to placebo and have a positive effect on child and adolescent PWS eating and repetitive behaviors. Additional knowledge of OXT's ability to reduce overeating could lead to improvement of patient's quality of life and physical health and reduction in familial stress.

The investigators propose a randomized double-blind 8 week treatment trial of intranasal OXT vs. placebo in 24 subjects aged 5 to 18 years with PWS in order to assess IN-OXT's affect on (1) Eating behaviors (2) Repetitive and disruptive behaviors and (3) Salivary OXT levels. If superior to placebo, this data will add to the current knowledge that OXT is an effective treatment for hyperphagia as well as other problematic symptomatology of PWS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female child outpatients aged 5 to 18 years
2. Diagnosis of PWS confirmed by genetic testing and patient medical records and history
3. Stable pharmacologic, educational, behavioral and/or dietary interventions for 4 weeks prior to the study start, and for the duration of the study.
4. Have a physical exam and laboratory results that are within the norms for PWS
5. Have a parent/caregiver/guardian that is able to consent for their participation and complete assessments regarding the child's development and behavior improvement throughout the study.

Exclusion Criteria:

1. Exposure to any investigational agent in the 30 days prior to randomization
2. Prior chronic treatment with oxytocin.
3. A primary psychiatric diagnosis other than ASD, including bipolar disorder, psychosis, schizophrenia, PTSD or major depressive disorder. These patients will be excluded due to potential confounding results.
4. Pregnant or lactating patients. IN-OXT has not been studied in pregnant or lactating women.
5. A medical condition that might interfere with the conduct of the study, confound interpretation of study results or endanger their own well-being.
6. Plan to initiate or change nonpharmacologic or pharmacologic interventions during the course of the study.
7. Females using an estrogen-based contraceptive. As an alternative to an estrogen based contraceptive, subjects will be counseled to use progesterone-based contraceptives; cervical caps; cervical sponges; or spermicidal foam in combination with a condom. Subjects will need to use a double barrier method to be in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- See also: Foundation for Prader Willi Research — http://www.fpwr.org/therapeutics-in-development-for-pws/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Oxytocin | Matched Placebo
Started | 11 | 12
Completed | 10 | 11
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin | Matched Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.72 (3.5) | 8.08 (3.82) | 8.87 (3.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 141.65 (15.23) | 124.91 (31.71) | 132.92 (26.11)
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 42.13 (14.6) | 38.53 (20.97) | 40.25 (17.89)
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.61 (5.04) | 21.2 (6.05) | 20.92 (5.47)
Hyperphagia Questionnaire (HQ)-Total [Mean (Standard Deviation); unit: score on a scale] | 27.91 (10.77) | 30.58 (8.08) | 29.3 (9.34)

OUTCOME MEASURES:

1. Primary Outcome: Hyperphagia Questionnaire (HQ)- Total Score
Description: The Hyperphagia Questionnaire (HQ)- Total Score. The HQ is a 11-item clinician-rated instrument that was designed to measure food related behaviors in PWS. Items map onto 3 subscales; Hyperphagic Behavior, Hyperphagic Drive, and Hyperphagia Severity. The subscales are summed together to compute the Total Score. The Total Score ranges from 11-55, with higher scores indicating more hyperphagia and a worse outcome.
Time Frame: Assessed trends over multiple time points (weeks 0, 2, 4, 6, and 8), week 0 (baseline), week 4 and week 8 are reported.
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 27.91 (10.77) | 30.58 (8.08)
  Week 4: number analyzed (Participants) | 10 | 9
  Week 4 | 27.4 (9.85) | 23.33 (8.41)
  Week 8: number analyzed (Participants) | 11 | 11
  Week 8 | 26.91 (11.67) | 25.09 (9.86)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.059, Mixed effects model — Mixed effects model with random slopes and intercepts, including main effects for time and treatment group and a time by treatment interaction term

2. Primary Outcome: Hyperphagia Questionnaire (HQ)- Behavior Factor Score
Description: The Hyperphagia Questionnaire (HQ)- Behavior Factor Score assesses food seeking behaviors (e.g., stealing food). The Behavior Factor Score ranges from 5-25, with higher scores indicating more hyperphagic behaviors and a worse outcome.
Time Frame: Assessed trends over multiple time points (weeks 0, 2, 4, 6, and 8), week 0 (baseline), week 4 and week 8 are reported.
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 9.55 (5.01) | 9.75 (3.47)
  Week 4: number analyzed (Participants) | 10 | 9
  Week 4 | 9.4 (4.27) | 7.22 (2.64)
  Week 8: number analyzed (Participants) | 11 | 11
  Week 8 | 9.64 (4.9) | 8.09 (4.25)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.088, Mixed effects model — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Hyperphagia Questionnaire (HQ)- Drive Factor Score
Description: The Hyperphagia Questionnaire (HQ)- Drive Factor Score assesses the persistence in asking for food. The Drive Factor Score ranges from 4-20, with higher scores indicating higher hyperphagic drive and a worse outcome
Time Frame: Assessed trends over multiple time points (weeks 0, 2, 4, 6, and 8), week 0 (baseline), week 4 and week 8 are reported.
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 10.82 (4.81) | 13.58 (4.44)
  Week 4: number analyzed (Participants) | 10 | 9
  Week 4 | 11 (4.03) | 10.44 (5.46)
  Week 8: number analyzed (Participants) | 11 | 11
  Week 8 | 10.36 (4.84) | 10.55 (4.48)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.027, Mixed effects model; Mixed effects model with random slopes and intercepts, including main effects for time and treatment group and a time by treatment interaction term

4. Primary Outcome: Hyperphagia Questionnaire (HQ) -Severity Factor Score
Description: The Hyperphagia Questionnaire (HQ)- Severity Factor Score assesses the severity of hyperphagia. The Severity Factor Score ranges from 2-10, with higher scores indicating higher severity.
Time Frame: Assessed trends over multiple time points (weeks 0, 2, 4, 6, and 8), week 0 (baseline), week 4 and week 8 are reported.
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin (IN-OXT) | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 7.55 (2.62) | 7.25 (2.09)
  Week 4: number analyzed (Participants) | 10 | 9
  Week 4 | 7.00 (2.54) | 5.67 (2.45)
  Week 8: number analyzed (Participants) | 11 | 11
  Week 8 | 6.91 (2.74) | 6.45 (2.54)
Statistical Analysis 1: Comparison: Intranasal Oxytocin (IN-OXT) vs Matched Placebo; Test type: Superiority — Mixed effects model with random slopes and intercepts, including main effects for time and treatment group and a time by treatment interaction term; p = 0.16, Mixed effects model

5. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R) Ritualistic Behavior Factor Score
Description: The Repetitive Behavior Scale-Revised (RBS-R) Ritualistic Behavior Factor Score assesses ritualistic behaviors. Scores range from 0-18, with higher scores indicating more ritualistic behaviors and a worse outcome.
Time Frame: Trends over multiple time points (Weeks 0, 4, and 8).
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 6.27 (3.74) | 9.42 (5.00)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 4.50 (3.84) | 6.27 (3.77)
  Week 8: number analyzed (Participants) | 10 | 11
  Week 8 | 4.90 (3.73) | 6.64 (4.65)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.69, Mixed effects model; [statistical method as in outcome 3, analysis 1]

6. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R) Sameness Factor Score
Description: The Repetitive Behavior Scale-Revised (RBS-R) Sameness Factor Score assesses the need for sameness in the environment. Scores range from 0-33, with higher scores indicating more need for sameness and a worse outcome.
Time Frame: Trends over multiple time points (Weeks 0, 4, and 8).
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 9.36 (4.72) | 14.17 (8.07)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 6.6 (5.25) | 8 (6.6)
  Week 8: number analyzed (Participants) | 10 | 11
  Week 8 | 7.3 (5.17) | 7.55 (7.39)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.034, Mixed effects model — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R) Stereotyped Behavior Factor Score
Description: The Repetitive Behavior Scale-Revised (RBS-R) Stereotyped Behavior Factor Score assesses stereotyped behaviors. Scores range from 0-18, with higher scores indicating more stereotyped behaviors and a worse outcome.
Time Frame: Trends over multiple time points (Weeks 0, 4, and 8).
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 2.18 (2.52) | 3.33 (2.84)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 2.5 (3.76) | 2 (2.53)
  Week 8: number analyzed (Participants) | 10 | 11
  Week 8 | 2.2 (3.01) | 1.09 (1.58)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.009, Mixed effects model; [statistical method as in outcome 3, analysis 1]

8. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R) Compulsive Behavior Factor Score
Description: The Repetitive Behavior Scale-Revised (RBS-R) Compulsive Behavior Factor Score assesses compulsive behaviors. Scores range from 0-24, with higher scores indicating more compulsive behaviors and a worse outcome.
Time Frame: Trends over multiple time points (Weeks 0, 4, and 8).
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 5.18 (6.9) | 7.5 (4.89)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 4.9 (5.69) | 5.27 (5.24)
  Week 8: number analyzed (Participants) | 10 | 11
  Week 8 | 4.5 (5.99) | 5.09 (5.41)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.033, Mixed effects model; [statistical method as in outcome 3, analysis 1]

9. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R) Self-Injurious Factor Score
Description: The Repetitive Behavior Scale-Revised (RBS-R) Self-Injurious Factor Score assesses self-injurious behaviors. Scores range from 0-24, with higher scores indicating more self-injurious behaviors and a worse outcome.
Time Frame: Trends over multiple time points (Weeks 0, 4, and 8).
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 5.00 (2.97) | 2.82 (2.86)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 4.40 (2.76) | 3.45 (5.68)
  Week 8: number analyzed (Participants) | 10 | 11
  Week 8 | 4.40 (2.46) | 3.36 (5.78)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.78, Mixed effects model; [statistical method as in outcome 3, analysis 1]

10. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R) Restricted Interest Factor Score
Description: The Repetitive Behavior Scale-Revised (RBS-R) Restricted Interest Factor Score assesses restricted interests. Scores range from 0-12, with higher scores indicating more restricted interests and a worse outcome.
Time Frame: Trends over multiple time points (Weeks 0, 4, and 8).
Population: 1 subject discontinued oxytocin early and 1 subject discontinued placebo early
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intranasal Oxytocin | Matched Placebo
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 3.27 (3.55) | 5.17 (3.27)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 2.20 (1.81) | 4.00 (3.13)
  Week 8: number analyzed (Participants) | 10 | 11
  Week 8 | 2.10 (2.13) | 3.73 (3.82)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Matched Placebo; Test type: Superiority; p = 0.53, Mixed effects model; [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Intranasal Oxytocin (IN-OXT) | Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 7/11 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Oxytocin (IN-OXT) (N=11) | Matched Placebo (N=12)
Fatigue (General disorders) | 2 (2) | 2 (2)
Increased Thirst (General disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Increased cataplexy (Nervous system disorders) | 1 (1) | 0 (0)
Increased movements, involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (nose bleed) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (3) | 1 (1)
Scraped Knee (General disorders) | 1 (1) | 0 (0)
Stomach Virus (General disorders) | 0 (0) | 1 (1)
Altitute Sickness (General disorders) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis Infective (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Otitis (Infections and infestations) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Worsening eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No